CLINICAL TRIAL: NCT00352183
Title: A Multicenter, Double-Blind, Randomized Study to Compare the Efficacy and Safety of the Combination of 145 mg Fenofibrate and 40 mg Simvastatin With 40 mg Simvastatin Monotherapy in Patients With Mixed Dyslipidemia at Risk of Cardiovascular Disease Not Adequately Controlled by 40 mg Simvastatin Alone.
Brief Title: Comparison of the Combination of Fenofibrate and 40 mg Simvastatin Versus 40 mg Simvastatin Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Martine Guy, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C LF0242780-01 05 02; ACTRN012605000777695
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Cardiovascular Diseases
Keywords: Hyperlipidemia Combined; Combination of fenofibrate and simvastatin
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fenofibrate; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Fenofibrate/Simvastatin
- 2 (Active Comparator)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Fenofibrate/Simvastatin — Combination of Fenofibrate and Simvastatin 40mg
  Arms: 1
Drug: Simvastatin — Simvastatin 40mg
  Arms: 2

SUMMARY:
Mixed or combined hyperlipidemia is a common metabolic disorder characterized by both hypercholesterolemia and hypertriglyceridemia. Statins and fibrates have complementary mechanisms and can be coadministered to patients with mixed hyperlipidemia. The overall objective of the study is to evaluate the efficacy and safety of combining fenofibrate and simvastatin in patients with mixed hyperlipidemia at risk of cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Mixed dyslipidemia

Exclusion Criteria:

* Diabetes,
* Known hypersensitivity to fenofibrate or simvastatin,
* Pregnant or lactating women,
* Contra-indication to fenofibrate or simvastatin,
* Unstable or severe cardiac disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2006-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Triglycerides | 12 weeks
Percent change from baseline to 12 weeks of treatment in HDL-C | 12 weeks
Percent change from baseline to 12 weeks of treatment in LDL-C | 12 weeks

SECONDARY OUTCOMES:
Percent change from baseline to 24 weeks of treatment in Triglycerides | 24 weeks
Percent change from baseline to 24 weeks of treatment in HDL-C | 24 weeks
Percent change from baseline to 24 weeks of treatment in LDL-C | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (67):
- Australia (25):
  - Site 204, Adelaide
  - Site 214, Adelaide
  - Site 203, Bendigo
  - Site 207, Brisbane
  - Site 208, Brisbane
  - Site 221, Brisbane
  - Site 202, Burnie
  - Site 201, Camperdown
  - Site 220, Coffs Harbour
  - Site 218, Daw Park
  - Site 212, Elizabeth Vale
  - Site 217, Fitzroy
  - Site 222, Fremantle
  - Site 216, Geelong
  - Site 225, Ingleburn
  - Site 213, Kippa-Ring
  - Site 209, Launceston
  - Site 219, Liverpool
  - Site 223, Malvern
  - Site 211, Meadowbrook
  - Site 224, Miranda
  - Site 210, Nambour
  - Site 205, Parkville
  - Site 206, Sale
  - Site 215, Sydney
- Estonia (7):
  - Site 301, Tallinn
  - Site 302, Tallinn
  - Site 303, Tallinn
  - Site 305, Tallinn
  - Site 306, Tallinn
  - Site 304, Tartu
  - Site 307, Tartu
- Hungary (10):
  - Site 603, Balatonfüred
  - Site 605, Budapest
  - Site 608, Budapest
  - Site 604, Gyöngyös
  - Site 602, Győr
  - Site 610, Hódmezővásárhely
  - Site 609, Kecskemét
  - Site 601, Miskolc
  - Site 607, Sopron
  - Site 606, Székesfehérvár
- Latvia (6):
  - Site 403, Daugavpils
  - Site 406, Jēkabpils
  - Site 401, Ogre
  - Site 402, Riga
  - Site 405, Riga
  - Site 404, Tukums
- Lithuania (8):
  - Site 502, Alytus
  - Site 503, Kaunas
  - Site 506, Kaunas
  - Site 505, Klaipėda
  - Site 507, Klaipėda
  - Site 508, Palanga
  - Site 504, Šiauliai
  - Site 501, Vilnius
- New Zealand (11):
  - Site 102, Auckland
  - Site 103, Auckland
  - Site 107, Blenheim
  - Site 101, Christchurch
  - Site 108, Dunedin
  - Site 104, Hamilton
  - Site 111, Hastings
  - Site 106, Nelson
  - Site 110, Newtown, Wellington
  - Site 109, Takapuna, Auckland
  - Site 105, Tauranga